CLINICAL TRIAL: NCT00214006
Title: Carotid Atherosclerotic Plaque Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0053
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
First, to establish a comparison of the pathophysiology of carotid atherosclerosis and the genetic and environmental variables that cause those plaques to become symptomatic. Second, to differentiate between vulnerable plaque and other types of plaque using ultrasound elastography, MRI data, trans-cranial doppler along with RF (radio frequency) analysis of back-scattered ultrasonic echoes.

DETAILED DESCRIPTION:
This is a multi-investigator study based on the pathophysiology of carotid atherosclerosis and the variables that cause certain plaques to become symptomatic.Patients enrolled in this study will be those patients undergoing a carotid endarterectomy. This will include both symptomatic and asymptomatic patients, and there are a variety of atherosclerotic risk factors representing this patient population.Patients may or may not have had strokes or transient ischemic attacks (TIAs).Pre-operatively patients will be reviewed for their medical history and atherosclerotic risk factors. Plaque removed during routine carotid endarterectomy will be examined for study purposes.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients aged 18-80 presenting for carotid endarterectomy

Exclusion Criteria:

* Patients not felt suitable for carotid endarterectomy and those with impaired decision-making capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing carotid endarectomy
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2001-11; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Lipid protein analysis and cognitive status comparison | 2008-2011
  Comparison studies will be done using the lipid protein analysis and imaging studies. The primary comparison will be between those that are symptomatic and those that are asymptomatic. Secondary comparisons will be done using the lipid protein analysis and patient history.
  Comparison of cognitive status between groups will be made using analysis of covariance in which the difference in follow-up score between groups (symptomatic/asymptomatic) is adjusted for baseline score. The baseline adjusted standard error is 6.4, which with 36 subjects per group will yield 90% power to detect a difference between groups of approximately 4.9 points at a significant level of 5%. We need 36 subjects per group to achieve the power stated. We have built in another 15% for projected dropout to insure we meet the final target.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Dempsey, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States